CLINICAL TRIAL: NCT07149467
Title: Ustekinumab and Upadacitinib for Induction and Maintenance Therapy in Patients With Refractory Crohn's Disease-A Multicenter, Randomized, Parallel-Controlled Study
Brief Title: Ustekinumab and Upadacitinib for Induction and Maintenance Therapy in Patients With Refractory Crohn's Disease: A Multicenter, Randomized, Parallel-Controlled Study
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiang Peng, Dr, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024ZSLYEC-312
Record Dates: First submitted 2025-08-24; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Crohn's Disease Aggravated; Crohn's Disease in Remission
Keywords: Crohn's Disease
MeSH Terms: interventions — Ustekinumab; upadacitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ustekinumab Group (Experimental): At Week 0:
  ≤55 kg: 260 mg administered by intravenous (IV) infusion.
  >55 kg and ≤85 kg: 390 mg administered by intravenous (IV) infusion.
  >85 kg: 520 mg administered by intravenous (IV) infusion.
  From Week 8 onward (i.e., at Week 8 and then every 8 weeks up to Week 52 or the end of the follow-up period):
  90 mg administered by subcutaneous (SC) injection.
  Interventions: Drug: Upadacitinib
- Upadacitinib Group (Active Comparator): From Week 0 to Week 12: 45 mg once daily, administered orally.
  From Week 13 through Week 52 or the end of the follow-up period: 30 mg once daily, administered orally.
  Interventions: Drug: Ustekinumab (approximately 6 mg/kg)

INTERVENTIONS:
Drug: Ustekinumab (approximately 6 mg/kg) — At Week 0:
  ≤55 kg: 260 mg administered by intravenous (IV) infusion.
  >55 kg and ≤85 kg: 390 mg administered by intravenous (IV) infusion.
  >85 kg: 520 mg administered by intravenous (IV) infusion.
  From Week 8 onward (i.e., at Week 8 and then every 8 weeks up to Week 52 or the end of the follow-up period):
  90 mg administered by subcutaneous (SC) injection.
  Arms: Upadacitinib Group
Drug: Upadacitinib — From Week 0 to Week 12: 45 mg once daily, administered orally.
  From Week 13 through Week 52 or the end of the follow-up period: 30 mg once daily, administered orally.
  Arms: Ustekinumab Group

SUMMARY:
Crohn's disease is a chronic inflammatory bowel disorder characterized primarily by abdominal pain and diarrhea [1,2]. Conventional treatments include corticosteroids and immunosuppressants (such as azathioprine, mercaptopurine, and methotrexate) [2,3]. The introduction of anti-tumor necrosis factor-α (TNF-α) inhibitors, such as infliximab and adalimumab, has significantly improved outcomes for patients with Crohn's disease, reducing complications and hospitalization rates [4]. However, both infliximab and adalimumab may lead to primary or secondary failure due to various reasons, including immunogenicity [5]. Novel biologics and small molecule drugs, such as ustekinumab and upadacitinib, offer new hope for the treatment of refractory Crohn's disease patients.

Ustekinumab is a monoclonal antibody targeting the p40 subunit of human interleukin (IL)-12/23. In the UNITI-2 study, the clinical remission rate at week 8 was 40% in the ustekinumab group, significantly higher than the 20% observed in the placebo group [6]. In the STARDUST study, the clinical remission rate at week 16 reached 68% in biologic-naïve patients and remained as high as 65% even in patients who had failed prior biologic therapy [7]. Upadacitinib is an orally administered JAK1 inhibitor that has now been approved for Crohn's disease in our region. In the recent U-EXCEED study, which enrolled refractory Crohn's disease patients who had failed at least one prior biologic therapy, the clinical remission rate at week 12 was 38.9%, significantly higher than that of the placebo group [8]. However, there is a lack of active head-to-head studies comparing the efficacy and safety of these two novel agents.

Our objective is to evaluate the efficacy and safety of ustekinumab and upadacitinib in the treatment of refractory Crohn's disease, thereby providing a theoretical basis for clinicians and patients in making informed therapeutic decisions.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, regardless of gender;

Diagnosis of Crohn's disease for at least 3 months or more based on medical history, laboratory tests, endoscopy, and imaging, in accordance with the Chinese Consensus on Inflammatory Bowel Disease;

Presence of one or more ulcers (in the ileum or colon) during colonoscopy, with an SES-CD score of at least 3;

Current or previous failure or intolerance to at least one anti-TNF-α therapy (infliximab or adalimumab);

Subjects taking oral corticosteroids (e.g., prednisone) are allowed a prednisone equivalent dose of up to 40 mg/day, provided the dose has been stable for 3 weeks prior to baseline (Week 0) or documented discontinuation of these medications at least 3 weeks before baseline;

Subjects using anti-TNF-α agents (infliximab or adalimumab) must discontinue these drugs at least 8 weeks (for infliximab) or 4 weeks (for adalimumab) prior to baseline;

Meeting the following tuberculosis (TB) screening criteria:

1. No history of latent or active TB prior to screening, except for the following:

   Currently receiving treatment for latent TB without evidence of active TB (or starting treatment for latent TB before administration at Week 0);

   History of latent TB with evidence of adequate treatment completed within 5 years prior to the first dose of the study drug.

   The investigator should fully verify the prior TB treatment history and provide corresponding documentation.
2. No signs or symptoms suggestive of active TB based on medical history and/or physical examination;
3. No known recent close contact with an active TB patient, or if such contact has occurred, the subject should be referred to a TB specialist for additional evaluation and, if necessary, receive appropriate treatment for latent TB before or concurrently with the first dose of the study drug;
4. Within 2 months prior to the first dose of the study drug:

   A negative T-SPOT® test, or a newly positive T-SPOT® test with active TB excluded, and appropriate treatment for latent TB initiated before or concurrently with the first dose of the study drug. Subjects with an indeterminate initial T-SPOT® test result should undergo repeat testing. If the additional T-SPOT® test result remains persistently indeterminate, the subject should also start treatment for latent TB to be eligible for the study;
5. Within 3 months prior to the first dose of the study drug, a chest imaging examination performed by a qualified radiologist shows no evidence of current active TB or old inactive TB;

For female subjects, a negative pregnancy test confirmed before screening and strict contraception during the study period or postmenopausal status. Male subjects should practice strict contraception;

Signed informed consent form indicating that the subject understands the purpose of the study and the required procedures and is willing to participate in the study.

Exclusion Criteria:

* Crohn's disease potentially requiring surgery, or conditions that may affect the assessment of ustekinumab or upadacitinib treatment efficacy using CDAI, such as short bowel syndrome, severe or symptomatic strictures, or active stoma.

Current or suspected abscess. Recent cutaneous and perianal abscesses are not excluded if drained and adequately treated at least 3 weeks prior to baseline. Intra-abdominal abscesses are not excluded if drained and adequately treated at least 8 weeks before baseline and no further surgery is anticipated. Subjects with active fistulas may be included if no further surgery is expected and there is no current abscess.

Any form of intestinal resection or intra-abdominal surgery within 6 months prior to baseline, or hospitalization for intestinal obstruction within 3 months prior to baseline.

Use of any of the following medications or treatments within the specified timeframes before baseline:

1. Any other experimental drug for Crohn's disease, unless at least 3 months or 5 half-lives have passed since the last dose;
2. Intravenous corticosteroid therapy within 3 weeks prior to baseline;
3. Immunosuppressants such as azathioprine, 6-mercaptopurine, methotrexate, etc., within 4 weeks prior to baseline;
4. Plasmapheresis within 3 weeks prior to baseline.

Positive stool culture or test for other intestinal pathogens, including Clostridium difficile toxin, within 4 months before screening, unless repeated testing is negative and there are no signs of ongoing infection.

Receipt of BCG vaccine within 12 months before screening or any other live bacterial or viral vaccine within 2 weeks after baseline.

History of chronic or recurrent infectious diseases, including but not limited to chronic kidney infection, chronic chest infection, recurrent urinary tract infection, or infected skin wounds or ulcers.

Current signs or symptoms of infection, or recent history (within 8 weeks before baseline) of herpes zoster or serious infection (including any condition requiring hospitalization).

Evidence of current active infection on screening or any other available chest imaging, including tuberculosis, or nodules suspected to be pulmonary malignancy, unless confirmed by surgery or additional imaging with supporting documentation.

History of latent or active granulomatous infections, including histoplasmosis or coccidioidomycosis, before screening. For information on latent tuberculosis, refer to the inclusion criteria.

History of non-tuberculous mycobacterial infection or severe opportunistic infection.

Patients with viral hepatitis or HIV.

Comorbid diagnosis or any history of congestive heart failure or demyelinating disease.

Recent history of severe, progressive, or uncontrolled renal, hepatic, hematological, endocrine, pulmonary, cardiac, neurological, systemic lupus erythematosus, or psychiatric disorders.

History of organ transplantation (except corneal transplantation performed more than 3 months before screening).

Lymphoproliferative disorders (including lymphoma) or signs and symptoms suggestive of possible lymphoproliferative disease.

Known malignancy or history of malignancy.

Previous allergy immunotherapy for anaphylaxis prevention.

Inability or unwillingness to undergo multiple venipunctures due to poor tolerance or lack of easily accessible veins.

Known allergy, hypersensitivity, or intolerance to ustekinumab or upadacitinib or their excipients.

Clinically significant drug abuse issues (e.g., drugs or alcohol) at screening or within 12 months before baseline.

Current or planned participation in any other clinical study within the first 52 weeks of this study.

Any condition that, in the investigator's opinion, would make participation not in the subject's best interest or may prevent, limit, or confound the protocol-specified assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 454 (Estimated)
Dates: Start 2025-09-10 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
clinical remission rate | 16th week
  To compare the efficacy of ustekinumab versus upadacitinib in subjects with refractory Crohn's disease who had prior failure or intolerance to at least one anti-TNF-α therapy (infliximab or adalimumab), as assessed by the clinical remission rate at Week 16.

IPD SHARING:
Plan to Share IPD: No